CLINICAL TRIAL: NCT05131347
Title: Effects of a Motor Intervention Program on Motor Skills and Adaptive Functions for Children With Autism Spectrum Disorder
Brief Title: Effects of Motor Skill Occupational Therapy Intervention ON ASD (Motion ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Yi Lin, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-BR-109-011
Record Dates: First submitted 2021-10-28; First posted 2021-11-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; motor skills; adaptive functions
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor intervention (Experimental): Children in the motor intervention group will receive a 8-week motor intervention program. Each week will be of 1.5-hour duration.
  Interventions: Behavioral: motor intervention
- cognitive intervention (Active Comparator): Children in the cognitive intervention group will receive a 8-week cognitive training program. Each week will be of 1.5-hour duration.
  Interventions: Behavioral: cognitive intervention

INTERVENTIONS:
Behavioral: motor intervention — Children in the motor intervention group will receive motor skills training based on motor learning theory. Movement activities include playing on trampoline and tilt board, walking on knees, toes and heels, creeping and crawling under different obstacles, jumping forward and backward, driving scooter board, playing balance devices, hopping, and visual motor coordinated movement. These activities are designed from easy to complex.
  Arms: motor intervention
Behavioral: cognitive intervention — Children in the cognitive intervention group will receive cognitive training. The activities consist of 12 exercises with progressive cognitive demands at 10 levels to improve cognitive functions such as attention, cognitive flexibility, inhibitory control, and working memory.
  Arms: cognitive intervention

SUMMARY:
The study will be a randomized controlled trial, which will aim to establish the appropriate and feasible content of the planned motor intervention program. A sample of 30 young children with ASD (4 to 5 years old) will be randomly assigned to treatment and control groups. Children in the treatment group will receive a 8-week motor skill intervention program. Children in the control group will receive a 8-week cognitive training program. Each week will be of 1.5-hour duration. Outcome measurements will consist of the Bruininks-Oseretsky Test of Motor Proficiency-Second Edition Brief Form and Vineland Adaptive Behavior Scales-Third Edition. A two-factor mixed design ANOVA will be conducted to compare pre- and post-tests differences in the treatment and control groups. The findings of the proposed study will be useful for occupational therapists and clinicians to assist caregivers in implementing the intervention program and will contribute to knowledge regarding the effects of motor intervention program on increasing the motor skills of young children with ASD in Taiwan. Practitioners can design a standard treatment manual and provide information for implementing the motor intervention program. The expected results will help clinicians apply empirical knowledge to provide and promote the health and development of young children with ASD.

DETAILED DESCRIPTION:
Introduction: Preschool children with autism spectrum disorder may have motor difficulties in performing daily activities. Therefore, effective and economical interventions are very important to support them. However, the empirical evidence was still weak due to poor research designs and little research was comprehensively investigated children's motor performance. Aim: This study will implement a dose-matched control group and comprehensive measurements to examine if the motor skill intervention program will improve children's motor performance. Hypotheses: The hypothesis will be that the better improvements would show in the motor skill intervention program than those in the cognitive training program. Method: Thirty preschool children with autism spectrum disorder will be recruited and randomly assigned to either the motor skill intervention program group or the cognitive training program group after pretest phase. Both groups will conduct 8-week intervention programs and be assessed after interventions. Children's motor performance will be assessed by the Bruininks-Oseretsky Test of Motor Proficiency-Second Edition Brief Form and the Vineland Adaptive Behavior Scales.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ASD by registered pediatric psychiatrists according to the Diagnostic and Statistical Manual-5th Edition
* aged 48 to 71 months old
* had no sensory impairments, such as visual or hearing impairments

Exclusion Criteria:

* diagnosed with additional diseases, comorbidities, or presence of other disorders, such as epilepsy, attention deficit hyperactivity disorder (ADHD), or Fragile X syndrome
* children with physical disabilities caused by head injuries, or neurological disorders
* the inability to follow researcher's instructions and complete the research procedures

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) Brief Form | 8 weeks
  The Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) Brief Form uses a subtest and composite structure that highlights motor performance in the broad functional areas of stability, mobility, strength, coordination, and object manipulation. Scale scores (mean = 15, standard deviation = 5), confidence intervals, age equivalents, and descriptive categories are used to describe subtest performance. Standard scores (mean = 50, standard deviation = 10), confidence intervals, percentile ranks, and descriptive categories are used to describe motor performance. The higher the scores are, the better performance the children achieve.
Vineland Adaptive Behavior Scales-Third Edition | 8 weeks
  The Vineland Adaptive Behavior Scales-Third Edition (VABS-3) comprises four domains, that is, communication, daily living skills, socialization and motor skills, for assessing adaptive functioning in children aged 3 to 12 years old. The raw score in each domain and total raw score are converted to an age-equivalent score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The range for each subscale is from 20 to 140. The subscales are summed to compute a total score, ranging from 80 to 560. The higher the scores are, the better adaptive functioning the children achieve.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Yi Lin, ScD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsaedi RH. An Assessment of the Motor Performance Skills of Children with Autism Spectrum Disorder in the Gulf Region. Brain Sci. 2020 Sep 3;10(9):607. doi: 10.3390/brainsci10090607. PMID 32899306